CLINICAL TRIAL: NCT03466255
Title: Vascular Imaging as a Barometer for the Early Detection of Cardiovascular Disease
Brief Title: Early Detection of Cardiovascular Disease
Acronym: VIBE
Status: Completed | Type: Observational
Sponsor: Dr. Amer Johri (Other)
Collaborators: Lantheus Medical Imaging (Industry)
Responsible Party: Sponsor-Investigator, Dr. Amer Johri, Associate Professor, Queen's University
Organization: Queen's University (Other)
Other Study IDs: DMED-1927-16; CG#17006 (Other Grant/Funding Number: Lantheus Medical Imaging, Inc.); ER15-11-029 (Other Grant/Funding Number: Ministry of Research, Innovation and Science - Ontario)
Record Dates: First submitted 2018-02-27; First posted 2018-03-15 (Actual); Last update posted 2022-06-09 (Actual); Status verified 2022-06

CONDITIONS: Atheroma; Cardiac Disease; Vascular Diseases; Atherosclerosis; Myocardial Infarction; Acute Coronary Syndrome
MeSH Terms: conditions — Plaque, Atherosclerotic; Heart Diseases; Vascular Diseases; Atherosclerosis; Myocardial Infarction; Acute Coronary Syndrome | interventions — High-Energy Shock Waves

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cardiac outpatients: Subjects referred for outpatient coronary angiography.
  Interventions: Other: Ultrasound

INTERVENTIONS:
Other: Ultrasound — Contrast-enhanced ultrasound (CEUS)
  Other Names: Contrast injection - Definity(R)

SUMMARY:
The investigators plan to evaluate the correlation between carotid plaque enhancement on Contrast-enhanced ultrasound (CEUS), significant coronary artery disease (CAD), and cardiovascular (CV) outcomes in a systematic manner. The investigators hypothesize that increased levels of CEUS-detected vulnerable carotid plaque will be predictive of CV risk determined by angiography and future cardiovascular events.

DETAILED DESCRIPTION:
Study Design: The investigators will conduct a prospective, single-center, observational study at the Cardiovascular Imaging Network at Queen's (CINQ, www.CINQLab.com). This facility allows a CEUS protocol to be conducted on the same day as the angiogram. It is anticipated that 100 participants can be recruited per month with a total target enrolment of up to 1000 participants.

Objectives

1. To determine the test characteristics (sensitivity, specificity, negative/positive predictive values) of carotid plaque by CEUS (Definity(R)) for predicting significant CAD (≥50% stenosis) in participants referred for angiography
2. To determine the test characteristics (sensitivity, specificity, predictive values) of carotid plaque by CEUS for predicting future CV events, such as death, stroke, myocardial infarction, and cardiovascular interventions.

ELIGIBILITY:
Inclusion criteria:

1. >18 years of age
2. Outpatients referred for clinically indicated angiography for assessment of CAD
3. Low - Intermediate Framingham risk (<20%)
4. Absence of clinical contraindication to angiography
5. Able and willing to give informed consent

Exclusion criteria:

1. Patients presenting with acute coronary syndrome
2. Patients with previously known significant CAD (any lesion >50%) or percutaneous coronary intervention or coronary artery bypass surgery
3. Previous carotid surgery or angioplasty
4. Documented allergy to echo contrast

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects referred for outpatient coronary angiography will be screened for inclusion.
Sampling Method: Non-Probability Sample
Enrollment: 610 (Actual)
Dates: Start 2016-12-06 (Actual); Primary Completion 2021-06-08 (Actual); Study Completion 2022-01-11 (Actual)

PRIMARY OUTCOMES:
Maximum Plaque Height (physiological parameter) | 4 years
  Caliper measurement of carotid plaque height on ultrasound images, using GE EchoPAC software. The maximum height of either side will be used to correlate to severity of angiographic CAD and neovascularization score.
Total Plaque Area (physiological parameter) | 4 years
  Area measurement of carotid plaque on ultrasound images (right + left side), using GE EchoPAC software. The total plaque area will be used to correlate to severity of angiographic CAD and neovascularization score.
Neovascularization (contrast enhancement intensity) (physiological parameter) | 4 years
  A neovascularization score will be used to grade the "activity" of the carotid plaque per participants and be correlated to angiographic CAD, visualized and manually counted using GE EchoPAC software.
Contrast wash-in time (physiological parameter) | 4 years
  Time of contrast entering the plaque will be assessed to see if it correlates to severity of angiographic CAD, using GE EchoPAC software.

SECONDARY OUTCOMES:
Participants CV outcome follow-up (data linkage through the Institute for Clinical Evaluative Sciences: ICES) | 5 years
  Participants will be followed for major adverse cardiac event over 5 years. Number of events will be correlated to carotid plaque measurements.

CONTACTS AND LOCATIONS:
Overall Officials: Amer M Johri, MD, Principal Investigator — Queen's University
Locations (1):
- Queen's University, Cardiovascular Imaging Network at Queen's (CINQ), Kingston General Hospital, Kingston, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Cardiovascular Imaging Network at Queen's — http://www.cinqlab.com